CLINICAL TRIAL: NCT03807336
Title: Improving Outcome for Children Through Treatment of Their Parents - Comparing Emotion-Focused Parent Skills Training With Emotion Coaching Parent Program for Children With Externalizing and Internalizing Symptoms: a Randomized Controlled Trial
Brief Title: Clinical Trial of Emotion-Focused Skills Training for Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institutt for Psykologisk Radgivning (Other)
Collaborators: University of Oslo (Other); The Research Council of Norway (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nadia_RCT_2018
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: F01.318 Child Rearing; F01.470 Emotions; F01.145.179 Child Behavior

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiential Condition (Experimental): This group will receive an experiential version of the program Emotion-Focused Skills Training for Parents, meaning they will engage in tasks that are supposed to activate the parents emotional system, providing them with a deeper sense of understanding towards their child.
  Interventions: Behavioral: Emotion-Focused Skills Training for Parents - Experiential; Behavioral: Emotion-Focused Skills Training for Parents - Psychoeducational
- Psychoeducational version (Active Comparator): This group will receive a non-experiential, psychoeducational version of the program Emotion-Focused Skills Training for Parents, meaning they will not engage in tasks that are meant to activate the parents emotional system.
  Interventions: Behavioral: Emotion-Focused Skills Training for Parents - Experiential; Behavioral: Emotion-Focused Skills Training for Parents - Psychoeducational

INTERVENTIONS:
Behavioral: Emotion-Focused Skills Training for Parents - Experiential — The intervention consists of a 2-day work shop given in a group format, in addition to 6 hours of parent supervision within 6 weeks after the work shop.
Behavioral: Emotion-Focused Skills Training for Parents - Psychoeducational — The intervention consists of a 2-day work shop given in a group format, in addition to 6 hours of parent supervision within 6 weeks after the work shop.

SUMMARY:
Children with externalizing and internalizing symptoms has been linked to poor emotional competence, problematic understanding and regulation of emotions. A number of recent studies demonstrates the importance of parents' active involvement in the child's recovery process and support the empirical relationship between parenting style and child symptoms. Emotional awareness and acceptance of painful emotional experience in parents leads to reduction in how these emotions are experienced in response to stressors in children. This makes the parent less vulnerable to rumination or suppression of negative emotional experience related to the child. In addition, it releases parents' emotional capacity to be mentally present and emotionally available for their child. Although neuro-affective principles from research have been incorporated in the therapeutic approaches for adults, there are currently no programs that target these mechanisms in working with children with mental health difficulties. Emotion Focused Skills Training (EFST) is an easily administrated, cost efficient treatment program specifically directed towards the parental role in promoting change in children. In this randomized controlled trial, we will compare experiential process oriented EFST with a psycho-educational version of EFST on parents of children aged 6-13 with externalizing or internalizing symptoms. Parents of 236 children will receive a two days course and 6 hours of individually delivered treatment within a 10 weeks period, either with the experiential version of EFST or the psycho-educational version. Feedback regarding outcome on externalizing and internalizing problems will be obtained from parents and teachers at 5 different periods: baseline, treatment completion and at 3, 6 and 9 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children between 6-13 with either internalizing problems, externalizing problems, or both.
* An overall final assessment of whether it is likely that the parents will be able to fully participate in the study.
* Parents who live with the child at least 50% of the time.
* Parents who agree that they need help and are motivated for the treatment.
* Parents and children who speak Norwegian
* Parents who have the time to participate in the intervention program.
* Parents who are willing to collaborate with the childs school and contact with the school teacher.

Exclusion Criteria:

* Parents: Serious or chronic mental health difficulties such as psychosis, bipolar disorder, organic disorder, ongoing substance abuse, do.
* documented sexual abuse, serious mental health problems, organic disorder and/or disability in the child.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Change in SDQ-P 4-17 - Strengths and Difficulties Questionnaire and impact supplement for the parents of 4-17 year olds All 5 subscales and total score will be used. | Pre, post (0 months after completed intervention), 3, 6 and 9 months follow up
Change in ASEBA Child Behavior Checklist for Ages 6-18 All eight subscales and total scores will be used. | Pre, post (0 months after completed intervention), 3, 6 and 9 months follow up
Change in ASEBA - Child Behavior Checklist - Teacher Report Form All eight subscales and total scores will be used. | Pre, post (0 months after completed intervention), 3, 6 and 9 months follow up

SECONDARY OUTCOMES:
Outcome Questionnaire 45, Version 2, for the parents | Pre, post (0 months after completed intervention), 3, 6 and 9 months follow up
  Outcome questionnaire designed to evaluate a psychotherapy client's progress initially and throughout treatment.
Difficulties in Emotion Regulation Scale | Pre, post, 3 months, 6 months, 9 monthsPre, post (0 months after completed intervention), 3, 6 and 9 months follow up
Forms of Self-Criticising/Attacking & Self-Reassuring Scale All 3 subscales will be used: Inadequate self, Hated self, Reassured self. | Pre, post (0 months after completed intervention), 3, 6 and 9 months follow up

OTHER OUTCOMES:
Parents Beliefs About Children's Emotions questionnaire Full scale | Pre, post (0 months after completed intervention), 3, 6 and 9 months follow up
Parents Sense of Competence Scale Full scale | Pre, post (0 months after completed intervention), 3, 6 and 9 months follow up
Coping with Children's Negative Emotion Scale Full scale | Pre, post (0 months after completed intervention), 3, 6 and 9 months follow up
Affect Integration Inventory Full scale: global affect integration | Pre, post (0 months after completed intervention), 3, 6 and 9 months follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Institutt for Psykologisk rådgivning, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ansar N, Nissen Lie HA, Stiegler JR. The effects of emotion-focused skills training on parental mental health, emotion regulation and self-efficacy: Mediating processes between parents and children. Psychother Res. 2024 Apr;34(4):518-537. doi: 10.1080/10503307.2023.2218539. Epub 2023 Jun 13. PMID 37311111